CLINICAL TRIAL: NCT00679289
Title: Phase II Study of the Anti-Ganglioside GD3 Mouse/Human Chimeric Antibody KW2871 Combined With High Dose Interferon-α2b in Patients With Metastatic Melanoma
Brief Title: Phase II Study of KW2871 Combined With High Dose Interferon-α2b in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: University of Pittsburgh (Other); University of Chicago (Other); Life Science Pharmaceuticals (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUD2007-001; UPCI07-023; UCH15689B
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Results first posted 2018-02-09 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Metastatic Melanoma; Cutaneous Melanoma
Keywords: KW2871; Ecromeximab; Anti-ganglioside; Antibody; Interferon alpha; Metastatic melanoma
MeSH Terms: conditions — Melanoma | interventions — Introns; ecromeximab

STUDY DESIGN:
Intervention Model Description: Dose-escalation cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): KW2871: 5 mg/m^2 IV every 2 weeks until disease progression
  HDI: 20 MU/m^2 IV QD for 5 days/week for 4 weeks, then 10 MU/m^2 SC 3 days/week until disease progression
  Interventions: Drug: HDI; Drug: KW2871
- Cohort 2 (Experimental): KW2871: 10 mg/m^2 IV every 2 weeks until disease progression
  HDI: 20 MU/m^2 IV QD for 5 days/week for 4 weeks, then 10 MU/m^2 SC 3 days/week until disease progression
  Interventions: Drug: HDI; Drug: KW2871
- Cohort 3 (Experimental): KW2871: 20 mg/m^2 IV every 2 weeks until disease progression
  HDI: 20 MU/m^2 IV QD for 5 days/week for 4 weeks, then 10 MU/m^2 SC 3 days/week until disease progression
  Interventions: Drug: HDI; Drug: KW2871

INTERVENTIONS:
Drug: HDI — 20 MU/m^2 IV QD for 5 days/week for 4 weeks, then 10 MU/m^2 SC 3 days/week until disease progression
  Other Names: Interferon-α2b; Intron A
Drug: KW2871 — 5 mg/m^2 IV every 2 weeks until disease progression
  Other Names: Ecromeximab
  Arms: Cohort 1
Drug: KW2871 — 10 mg/m^2 IV every 2 weeks until disease progression
  Other Names: Ecromeximab
  Arms: Cohort 2
Drug: KW2871 — 20 mg/m^2 IV every 2 weeks until disease progression
  Other Names: Ecromeximab
  Arms: Cohort 3

SUMMARY:
This was a Phase 2, open-label study of KW2871 (ecromeximab) in combination with high-dose interferon-α2b (HDI) in patients with metastatic melanoma. The primary objectives of this study were to assess progression-free survival (PFS) and safety. The secondary objectives were to assess the objective response rate, KW2871 pharmacokinetics (PK), and other exploratory immunology as indicated (e.g., development of human anti-chimeric antibodies [HACA], activity of antibody-dependent cell-mediated cytotoxicity [ADCC] and complement-dependent cytotoxicity [CDC] in peripheral blood, number and functional state of tumor-infiltrating immune cells and expression of GD3 in immune and tumor cells of tumor biopsies, and markers of interferon [IFN] response/resistance and markers of resistance to ADCC/CDC in peripheral blood mononuclear cells [PBMCs]).

DETAILED DESCRIPTION:
Eligible patients were sequentially enrolled into dose-escalating cohorts to receive KW2871 intravenously (IV) once every 2 weeks starting on Day 3 of Week 1 at the following doses: 5 mg/m^2 in Cohort 1, 10 mg/m^2 in Cohort 2, and 20 mg/m^2 in Cohort 3. HDI was administered concurrently at a dose of 20 million units (MU)/m^2 IV once daily (QD) for 5 consecutive days per week for 4 weeks (induction phase), followed by 10 MU/m^2 administered subcutaneously (SC) 3 times per week (maintenance phase). Patients received KW2871 and HDI combination therapy until disease progression requiring treatment intervention that would have interfered with the interpretation of the study results.

Initially, 3 patients were enrolled within a cohort and evaluated for dose-limiting toxicity (DLT) and regimen-limiting toxicity (RLT) for the first 8 weeks of study treatment. If 1 of 3 patients experienced an RLT, the cohort was expanded to 6 patients. Escalation to the next higher dose cohort proceeded if the RLT rate was <33% (0/3 or 1/6 patients) in a given cohort. The combination treatment was considered safe if ≤ 20% patients experienced RLT.

DLT was defined as any adverse event (AE) that required reduction of the HDI dose or discontinuation of KW2871. RLT was defined as an HDI-related DLT that required more than 2 dose reductions of HDI during the induction phase or the first 4 weeks of the maintenance phase, or any KW2871- or regimen-related DLT.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age.
2. Histologically proven metastatic cutaneous, mucosal, or unknown primary melanoma.
3. Measurable disease using Response Evaluation Criteria in Solid Tumors (RECIST).
4. Ambulatory (Eastern Cooperative Oncology Group [ECOG] performance status 0 or 1) or expected survival ≥ 4 months.
5. Within the last 2 weeks prior to study day 1, the following laboratory parameters within the ranges specified:

   * Hemoglobin: ≥ 9 g/dL
   * Platelets: ≥ 100 x 10^9/L
   * Neutrophils: ≥ 1.5 x 10^9/L
   * International normalized ratio: ≤ 2.0 (≤ 3.0 if on warfarin therapy)
   * Serum creatinine: ≤ 1.5 x upper limit of normal (ULN)
   * Serum total bilirubin: ≤ 1.5 x ULN
   * Aspartate aminotransferase/alanine aminotransferase: ≤ 2.5 x ULN
6. Able and willing to give valid written informed consent.

Exclusion Criteria:

1. Other malignancy within 3 years prior to study entry for which the patient received active treatment, except for treated melanoma or non-melanoma skin cancer, cervical cancer, and breast carcinoma in situ.
2. Mental impairment that may have compromised the ability to give informed consent and comply with the study requirements.
3. Participation in any other clinical trial involving chemotherapy, radiotherapy, or other immunotherapy within 4 weeks prior to study enrollment.
4. Prior exposure to anti-GD3 antibodies.
5. Pregnancy or breastfeeding.
6. Women of childbearing potential who refused or were unable to use effective means of contraception.
7. Active autoimmune or other disorders that required systemic treatment with immunomodulatory or immunosuppressant medications (i.e., corticosteroids, cyclophosphamide, methotrexate, other biologics). Corticosteroids at substitution doses were allowed.
8. Metastatic brain disease was allowed provided that appropriate treatment had been administered (surgery or irradiation) and 2-month follow-up by brain magnetic resonance imaging (MRI) showed disease control (stability or regression).
9. Autoimmune-related hypothyroidism and vitiligo-like depigmentation were allowed provided the patient was medically stable with treatment (thyroid-hormone replacement or observation).
10. Serious medical illness, such as cardiovascular disease (uncontrolled congestive heart failure or hypertension, active ischemic disease of the heart [angina], recent [<3 months] myocardial infarction, severe cardiac arrhythmia), bleeding disorders, obstructive or restrictive pulmonary diseases, active systemic infections requiring antibiotics, serious intercurrent illness requiring hospitalization, inflammatory bowel disorders, or significant psychiatric disease, which in the opinion of the principal investigator would have prevented adequate informed consent or rendered study treatment unsafe or contraindicated.
11. Patients with clinical suspicion of human immunodeficiency virus (HIV) or hepatitis underwent the following viral tests: patients with HIV must have had negative antibodies; patients with hepatitis B virus must have had negative antigens; patients with hepatitis C virus must have had a negative test for serum antibodies. If any of the tests were positive, patients were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-03-28 (Actual); Primary Completion 2014-02-03 (Actual); Study Completion 2014-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M. Kirkwood, MD, Study Chair — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Chicago Hospital, Chicago, Illinois
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tarhini AA, Moschos SJ, Lin Y, Lin HM, Sander C, Yin Y, Venhaus R, Gajewski TF, Kirkwood JM. Safety and efficacy of the antiganglioside GD3 antibody ecromeximab (KW2871) combined with high-dose interferon-alpha2b in patients with metastatic melanoma. Melanoma Res. 2017 Aug;27(4):342-350. doi: 10.1097/CMR.0000000000000353. PMID 28489678
- See also: Abstract with option to purchase full text — http://journals.lww.com/melanomaresearch/Abstract/2017/08000/Safety_and_efficacy_of_the_antiganglioside_GD3.8.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: KW2871: 5 mg/m^2 IV every 2 weeks
  HDI: 20 MU/m^2 IV QD for 5 days/week for 4 weeks, then 10 MU/m^2 SC 3 days/week
- Cohort 2: KW2871: 10 mg/m^2 IV every 2 weeks
  HDI: 20 MU/m^2 IV QD for 5 days/week for 4 weeks, then 10 MU/m^2 SC 3 days/week
- Cohort 3: KW2871: 20 mg/m^2 IV every 2 weeks
  HDI: 20 MU/m^2 IV QD for 5 days/week for 4 weeks, then 10 MU/m^2 SC 3 days/week
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started (Received at least 1 dose of KW2871 and initial treatment with HDI) | 6 | 6 | 24
Completed | 1 | 0 | 1
Not Completed | 5 | 6 | 23
Not completed — Progressive disease | 4 | 5 | 18
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Physician Decision | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (includes all patients who received at least 1 dose of KW2871 and initial treatment with HDI)
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 6 | 6 | 24 | 36
Age, Continuous [Median (Full Range); unit: years] | 55 [27 to 70] | 61 [31 to 73] | 54 [36 to 72] | 54 [27 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 13 | 18
  Male | 4 | 3 | 11 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 24 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 6 | 24 | 36
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 24 | 36
Body Mass Index [Median (Full Range); unit: kg/m^2] | 24.4 [20.7 to 26.5] | 29.4 [27.6 to 39.2] | 26.3 [18.3 to 45.9] | 26.5 [18.3 to 45.9]

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-free Survival (PFS) With 95% Confidence Intervals
Description: PFS was calculated from the date of the first infusion to the date of documented progression or death, whichever occurred first. PFS analyses were performed using Kaplan-Meier methods for all patients combined and for patients in Cohort 3. Based on published results from Phase 3 randomized clinical trials in patients with metastatic melanoma at the time of study initiation, 2.5 months was estimated as a conservative (i.e., somewhat high) external standard of median PFS. The intent of this study was to improve this standard by ≥ 70% to a median PFS of ≥ 4.3 months for patients treated with KW2871 combined with HDI. If the therapeutic target of 4.3 months for median PFS represented the true underlying treatment effect of KW2871 plus HDI, then 23 patients would provide 80% power to detect a statistically significant improvement (α = 0.05; 1-sided test) over the 2.5-month external standard.
Time Frame: From baseline through up to 17 months post-baseline
Population: Patients who received initial treatment with HDI and at least 1 infusion of KW2871 and experienced a PFS event (progression or death).
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Total: All evaluable patients in Cohorts 1, 2, and 3 combined
Arm/Group | Cohort 3 | Total
Number analyzed (Participants) | 24 | 34
months | 1.93 [1.00 to 3.80] | 2.53 [1.93 to 3.83]

2. Primary Outcome: Number of Patients With Treatment-emergent Adverse Events (TEAEs)
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0, as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (life-threatening), or Grade 5 (fatal). TEAEs were reported based on clinical laboratory tests, physical examinations, and vital signs from pre-treatment through the study period. Causal relationship of each TEAE to study treatment was evaluated by the investigator separately for HDI and KW2871. Regimen-limiting toxicity was defined as an HDI-related dose-limiting toxicity (DLT) that required more than 2 dose reductions of HDI during the induction phase or the first 4 weeks of the maintenance phase, or any KW2871- or regimen-related DLT.
Time Frame: From baseline through up to 17 months post-baseline
Population: Patients who received initial treatment with HDI and at least 1 infusion of KW2871.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 6 | 6 | 24
Participants
  Any TEAE | 6 | 6 | 24
  Maximum TEAE Severity Grade 1/2 | 0 | 1 | 2
  Maximum TEAE Severity Grade 3 | 5 | 2 | 20
  Maximum TEAE Severity Grade 4 | 1 | 2 | 1
  Maximum TEAE Severity Grade 5 | 0 | 1 | 1
  Any HDI-related TEAE | 6 | 6 | 24
  Any KW2871-related TEAE | 4 | 5 | 7
  Any SAE | 2 | 1 | 7
  Any TEAE leading to withdrawal of HDI+KW2871 | 0 | 1 | 3
  Any TEAE leading to withdrawal of HDI only | 0 | 0 | 1
  Any TEAE leading to withdrawal of KW2871 only | 0 | 0 | 1
  Regimen-limiting toxicity | 0 | 0 | 2

3. Secondary Outcome: Number of Patients With Best Overall Tumor Response
Description: Tumor responses were evaluated using whole body computed tomography and categorized according to the Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0) at Screening, on Days 29, 57, 85, 115, 143, 171, 227, 283, 339, and at the End of Study Visit. Patients who were treated beyond 49 weeks were to undergo clinical and radiologic assessments per the standard of care. Per RECIST, target lesions are categorized as follows: Complete Response (CR): Disappearance of all target lesions [no evidence of disease]; Partial Response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD): small changes that do not meet above criteria.
Time Frame: From baseline through up to 17 months post-baseline
Population: Patients who received initial treatment with HDI and at least 1 infusion of KW2871.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 6 | 6 | 24
Participants
  CR | 0 | 0 | 1
  PR | 1 | 0 | 0
  SD | 5 | 5 | 16
  PD | 0 | 1 | 7

4. Secondary Outcome: Number of Patients With Human Antichimeric Antibody (HACA) Reactivity To KW2871
Description: Blood samples were collected for the analysis of HACA at baseline, on Days 29, 115, 143, 171, 199, 227, 255, 283, 311, 339, and at the End of Study visit. Measurement of HACA development in plasma was performed with a BIAcore 2000 biosensor (Biacore AB, Uppsala, Sweden), using the BDF TM015 method. HACA positivity was defined as an increase in binding evident in the test channel but not in the control channel, with positivity assigned for values exceeding a uniform test threshold.
Time Frame: From baseline through up to 17 months post-baseline
Population: Patients who received initial treatment with HDI and at least 1 infusion of KW2871 and had at least 1 post-baseline plasma sample evaluated for HACA.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 6 | 6 | 16
Participants
  Baseline negative, post-baseline negative | 5 | 6 | 16
  Baseline negative, post-baseline positive | 1 | 0 | 0

5. Secondary Outcome: Maximum KW2871 Antibody Levels in Plasma Following the First Infusion
Description: Blood samples for pharmacokinetic (PK) measurements were collected at baseline and before and 30 minutes after the initial KW2871 infusion on Day 3. The KW2871 antibody protein in patient serum was measured using an enzyme-linked immunosorbent assay (ELISA). The lower limit of quantitation was determined to be 100 ng/mL.
Time Frame: At Baseline and Study Day 3
Population: Patients who received initial treatment with HDI and at least 1 infusion of KW2871 and had at least 1 plasma sample evaluated for KW2871 antibody levels.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 6 | 19
µg/mL | 3.22 (3.02) | 5.17 (5.07) | 9.18 (4.26)

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring between the signing of informed consent and the off-study date were documented, regardless of the causal relationship to study drug. AEs occurring after the first dose of study drug were considered treatment emergent (i.e., TEAEs). The AE reporting period for this study was up to 17 months.
Description: AE documentation included onset/resolution dates, severity using the NCI CTCAE (version 3.0), seriousness, study drug action taken, treatment, and outcome. Relationship to study drug was evaluated for both KW2871 and HDI. Treatment-related AEs included those with a "possible", "probable", or "definite" relationship to study drug; preferred terms were counted only once per patient at the maximum reported grade.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/6 | 1/24
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/6 | 7/24
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=6) | Cohort 3 (N=24)
Nausea (Gastrointestinal disorders) | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2
Hypotension (Vascular disorders) | 0 | 0 | 2
Appendicitis (Infections and infestations) | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=6) | Cohort 3 (N=24)
Chills (General disorders) | 6 | 6 | 22
Fatigue (General disorders) | 6 | 6 | 21
Pyrexia (General disorders) | 6 | 3 | 21
Oedema peripheral (General disorders) | 0 | 1 | 4
Pain (General disorders) | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 2
Axillary pain (General disorders) | 1 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0
Nodule (General disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 4 | 18
Vomiting (Gastrointestinal disorders) | 2 | 2 | 12
Constipation (Gastrointestinal disorders) | 2 | 2 | 12
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 11
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 3
Early satiety (Gastrointestinal disorders) | 0 | 0 | 3
Oral pain (Gastrointestinal disorders) | 0 | 0 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0
Gingival ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Lip pain (Gastrointestinal disorders) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 5 | 5 | 17
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 14
Dehydration (Metabolism and nutrition disorders) | 2 | 3 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 12
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 5 | 18
Gamma-glutamyltransferase increased (Investigations) | 3 | 4 | 17
Blood lactate dehydrogenase increased (Investigations) | 3 | 5 | 15
Alanine aminotransferase increased (Investigations) | 4 | 2 | 14
Haemoglobin decreased (Investigations) | 3 | 6 | 9
Blood creatine phosphokinase increased (Investigations) | 3 | 4 | 8
Weight decreased (Investigations) | 0 | 4 | 11
Blood alkaline phosphatase increased (Investigations) | 1 | 3 | 7
Platelet count decreased (Investigations) | 0 | 0 | 6
Lymphocyte count decreased (Investigations) | 0 | 0 | 4
Neutrophil count decreased (Investigations) | 0 | 0 | 3
Blood alkaline phosphatase (Investigations) | 0 | 1 | 1
International normalised ratio increased (Investigations) | 1 | 1 | 0
Neutrophil count (Investigations) | 0 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 2
Biopsy site unspecified abnormal (Investigations) | 1 | 0 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1
Blood calcium decreased (Investigations) | 0 | 0 | 1
Blood folate decreased (Investigations) | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 1 | 0
Body temperature fluctuation (Investigations) | 0 | 0 | 1
Breath sounds abnormal (Investigations) | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 1
Haemoglobin (Investigations) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0 | 0
Mean cell haemoglobin concentration decreased (Investigations) | 0 | 0 | 1
Monocyte count increased (Investigations) | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 1
Protein total decreased (Investigations) | 0 | 0 | 1
Protein total increased (Investigations) | 0 | 0 | 1
Red cell distribution width increased (Investigations) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 4 | 4 | 14
Neutropenia (Blood and lymphatic system disorders) | 4 | 5 | 13
Lymphopenia (Blood and lymphatic system disorders) | 2 | 1 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4 | 8
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 6
Haemoglobinaemia (Blood and lymphatic system disorders) | 0 | 0 | 5
Basophilia (Blood and lymphatic system disorders) | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Monocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 4 | 6 | 13
Headache (Nervous system disorders) | 4 | 3 | 11
Dizziness (Nervous system disorders) | 1 | 0 | 9
Nystagmus (Nervous system disorders) | 0 | 1 | 4
Tremor (Nervous system disorders) | 1 | 1 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 2
Anosmia (Nervous system disorders) | 0 | 1 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 1 | 7
Depression (Psychiatric disorders) | 2 | 2 | 5
Insomnia (Psychiatric disorders) | 3 | 0 | 4
Confusional state (Psychiatric disorders) | 0 | 0 | 4
Restlessness (Psychiatric disorders) | 0 | 0 | 4
Agitation (Psychiatric disorders) | 0 | 0 | 2
Delirium (Psychiatric disorders) | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 4
Exfoliative rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypocapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngeal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 2 | 3
Orthostatic hypotension (Vascular disorders) | 0 | 2 | 3
Hypertension (Vascular disorders) | 0 | 0 | 4
Haematoma (Vascular disorders) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 5
Candidiasis (Infections and infestations) | 2 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 1 | 2
Visual impairment (Eye disorders) | 0 | 0 | 2
Eye pruritus (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less